CLINICAL TRIAL: NCT01680237
Title: Cognitive Behavior Therapy vs Exposure in Vivo in the Treatment of Panic Disorder With Agoraphobia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Retirement of one of the PIs and participation in another multi center study, within which the same patient inclusion criteria were used.
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Dr. Tobias Teismann, Dr. Tobias Teismann, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BoSPmA
Record Dates: First submitted 2012-08-17; First posted 2012-09-07 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Panic Disorder With Agoraphobia
Keywords: cognitive behavior therapy; exposure in-vivo; panic disorder with agoraphobia
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavior therapy (Active Comparator): 1. Identification of bodily sensations, cognitions and safety behaviors characteristic of the individual patient
  2. Modification of dysfunctional beliefs and assumptions using socratic questioning and behavioral experiments
  3. Exposure in-vivo
  4. Relapse prevention
  Interventions: Behavioral: Cognitive behavior therapy
- Exposure in-vivo (Active Comparator): 1. Preparation of a brief behavior analysis of the individual case and construction of a hierarchy of relevant (internal and external) phobic situations
  2. Exposure with internal stimuli
  3. Exposure with external stimuli
  4. Relapse prevention
  Remark: In this condition there is no active work with the patient's catastrophic cognitions
  Interventions: Behavioral: Exposure in-vivo

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Treatment covers psychoeducation on the nature of anxiety and panic, interoceptive and intensified situational exposure exercises as well as identification and correction of maladaptive thoughts about anxiety and its consequences.
  Arms: Cognitive behavior therapy
Behavioral: Exposure in-vivo — Treatment covers psychoeducation on the nature of anxiety and panic, interoceptive and intensified situational exposure exercises.
  Arms: Exposure in-vivo

SUMMARY:
Panic disorder with agoraphobia is a prevalent and one of the most handicapping anxiety disorders. Although the efficacy of psychological treatment for panic disorder with agoraphobia has been the subject of a great deal of research, studies comparing cognitive-behavioral therapy and exposure in vivo have regularly been underpowered to detect small to moderate differences. Therefore, the primary purpose of the present study is to investigate if the combination of cognitive techniques with exposure in vivo is superior to the effects of exposure alone for patients with moderate to severe agoraphobia.

DETAILED DESCRIPTION:
Anxiety disorders are the most common group of mental illnesses, with lifetime prevalence estimates ranging between 10-30% (Kessler et al 2007). They are an economic burden on society and the sixth largest cause of disability globally (Baxter et al 2014; Fineberg et al 2013). Suffering from an anxiety disorder is distressing, with affected individuals reporting adverse effects on quality of life comparable to sufferers of major depressive disorder, and in excess of the population norm (Mendlowicz and Stein 2000). Panic disorder with agoraphobia is especially prevalent and one of the most handicapping anxiety disorders.

Although the efficacy of psychological treatment for panic disorder with agoraphobia has been the subject of a great deal of research (Sanchez-Meca, Rosa-Alcazar, Marin-Martinez & Gomez-Conesa, 2010), studies comparing cognitive-behavioral therapy and exposure in vivo have regularly been underpowered to detect small to moderate differences.

Therefore, the primary purpose of the present study is to investigate if the combination of cognitive techniques with exposure in vivo is superior to the effects of exposure alone for patients with moderate to severe agoraphobia. Participants suffering from panic disorder, agoraphobia receive exposure-based treatment with elements of cognitive restructuring (CBT-group) or without such elements (Exposure-only group) delivered according to treatment manuals and in individual sessions with a maximum of 30 sessions á 50 minutes. Both treatments cover psychoeducation on the nature of anxiety and panic, interoceptive and intensified situational exposure exercises. In the CBT group identification and correction of maladaptive thoughts about anxiety and its consequences is furthermore part of the treatment package.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of panic disorder with agoraphobia by trained clinician using a structured interview
* The anxiety disorder is considered to be the patient's main current problem
* Age between 18 and 65 years
* The patient has agreed to participate in the study

Exclusion Criteria:

- Diagnosis of bipolar disorder, psychotic disorder, alcohol/substance abuse or dependency (within past 3 months), prominent risk of self-harm, organic mental disorder; concurrent psychotherapeutic or psychopharmacological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-10; Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in the Mobility Inventory | 0, 6, 12 month after treatment
  Avoidance Behaviour

SECONDARY OUTCOMES:
Change (from baseline) in a Behavioral Approach Test | 0, 6, 12 month after treatment
  Participants are asked to go up a high and narrow church tower. The test yields number of floors (0-10) the patient achieves, recording the experienced anxiety level (0-100).

OTHER OUTCOMES:
Change (from baseline) in the Anxiety Disorder Interview Schedule | 0, 6, 12 month after treatment
  Remission Status

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Teismann, Dr., Principal Investigator — Ruhr-Universität Bochum
Locations (1):
- Zentrum für Psychotherapie, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Available upon request from August 2021
Access Criteria: Researchers in the field of anxiety disorders, meta-analysis, contact: tobias Teismann

REFERENCES:
- [Background] Sanchez-Meca J, Rosa-Alcazar AI, Marin-Martinez F, Gomez-Conesa A. Psychological treatment of panic disorder with or without agoraphobia: a meta-analysis. Clin Psychol Rev. 2010 Feb;30(1):37-50. doi: 10.1016/j.cpr.2009.08.011. PMID 19775792
- [Background] Kessler RC, Angermeyer M, Anthony JC, DE Graaf R, Demyttenaere K, Gasquet I, DE Girolamo G, Gluzman S, Gureje O, Haro JM, Kawakami N, Karam A, Levinson D, Medina Mora ME, Oakley Browne MA, Posada-Villa J, Stein DJ, Adley Tsang CH, Aguilar-Gaxiola S, Alonso J, Lee S, Heeringa S, Pennell BE, Berglund P, Gruber MJ, Petukhova M, Chatterji S, Ustun TB. Lifetime prevalence and age-of-onset distributions of mental disorders in the World Health Organization's World Mental Health Survey Initiative. World Psychiatry. 2007 Oct;6(3):168-76. PMID 18188442
- [Background] Baxter AJ, Vos T, Scott KM, Ferrari AJ, Whiteford HA. The global burden of anxiety disorders in 2010. Psychol Med. 2014 Aug;44(11):2363-74. doi: 10.1017/S0033291713003243. Epub 2014 Jan 22. PMID 24451993
- [Background] Fineberg NA, Haddad PM, Carpenter L, Gannon B, Sharpe R, Young AH, Joyce E, Rowe J, Wellsted D, Nutt DJ, Sahakian BJ. The size, burden and cost of disorders of the brain in the UK. J Psychopharmacol. 2013 Sep;27(9):761-70. doi: 10.1177/0269881113495118. Epub 2013 Jul 24. PMID 23884863
- [Background] Mendlowicz MV, Stein MB. Quality of life in individuals with anxiety disorders. Am J Psychiatry. 2000 May;157(5):669-82. doi: 10.1176/appi.ajp.157.5.669. PMID 10784456